CLINICAL TRIAL: NCT04387136
Title: Intraoperative Sublingual Sufentanil for Acute Pain in the Ambulatory Surgery Center
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANES-2020-28605
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Pain; Pain, Acute; Anesthesia
MeSH Terms: conditions — Pain; Acute Pain | interventions — Dsuvia; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublingual Sufentanil (Experimental): Participants in this arm will receive the intervention.
  Interventions: Drug: Sublingual Sufentanil
- Control (No Intervention): Participants in this arm will not receive an intervention.

INTERVENTIONS:
Drug: Sublingual Sufentanil — 15-30 minutes prior to planned emergence from anesthesia patients will either receive 30 mcg of sublingual sufentanil dispensed by the anesthesia provider.
  Other Names: Dsuvia; Sufenta
  Arms: Sublingual Sufentanil

SUMMARY:
The purpose of this study is to determine if a single dose of sublingual sufentanil given 15-30 minutes prior to wake up is efficacious at reducing recovery room time.

DETAILED DESCRIPTION:
This is a level I randomized prospective outcomes study comparing two groups of patients. Within 15-30 minutes of planned wake-up Group 1 will receive 30 mcg of sublingual sufentanil and group 2 will not receive sublingual sufentanil.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients undergoing outpatient ambulatory surgery undergoing general anesthesia for orthopedic surgery

Exclusion Criteria:

* non-english speaking patients
* patients who have allergy or intolerance to the study drugs or derivatives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Bern, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sublingual Sufentanil | Control
Started | 26 | 27
Completed | 25 | 25
Not Completed | 1 | 2
Not completed — Protocol Deviation by SOC staff | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sublingual Sufentanil | Control | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 14 | 18 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Initial Numeric Rating Scale (NRS) Pain Score Upon Arrival
Description: Pain is assessed on a scale of 0-10 (whole numbers). A score of 0 being no pain, 10 being maximum imaginable pain. Data collected upon arrival to Post-Anesthesia Care Unit (PACU).
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sublingual Sufentanil | Control
Number analyzed (Participants) | 25 | 25
score on a scale | 4 [0 to 6] | 4 [3 to 5]

2. Secondary Outcome: Opioid Use in Recovery Room
Description: Opioid medication type and dose will be recorded and converted to milligram morphine equivalents. Outcome is reported as the total milligram morphine equivalents of opioid medication used in the recovery room.
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: mg (morphine equivalent)
Arm/Group | Sublingual Sufentanil | Control
Number analyzed (Participants) | 25 | 25
mg (morphine equivalent) | 7.5 [0.0 to 22.5] | 15.0 [7.5 to 37.5]

3. Secondary Outcome: OBAS Score
Description: Overall Benefit of Analgesic Score (OBAS) is a 7-item multi-dimensional survey that assesses analgesia benefits. Items are scored on a scale from 0 (minimal) to 4 (maximal). Total score is a sum of the 7 item scores with question 7 scored as 4 minus the patient reported number. Total scores range from 0 to 28 with lower scores representing greater benefit from analgesic therapy.
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Sublingual Sufentanil | Control
Number analyzed (Participants) | 25 | 25
score | 1.0 [0.0 to 2.0] | 3.0 [1.0 to 3.0]

ADVERSE EVENTS:
Time Frame: 16 weeks from baseline
Arm/Group | Sublingual Sufentanil | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sublingual Sufentanil (N=25) | Control (N=25)
Anxiety (Psychiatric disorders) | 2 (3) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Post-operative nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT04387136/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04387136/ICF_001.pdf